CLINICAL TRIAL: NCT03318653
Title: Adherence to Blood Pressure Measurement Guidelines for Patients With End-stage Renal Disease on Renal Replacement Therapy (hæmodialysis or Peritoneal Dialysis)
Brief Title: Blood Pressure Measurement in Dialysed Patients
Acronym: DIALBP
Status: Completed | Type: Observational
Sponsor: PD Dr. Grégoire Wuerzner (Other)
Collaborators: University Hospital, Geneva (Other); Universitair Ziekenhuis Brussel (Other); Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other); Royal Infirmary of Edinburgh (Other); Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor-Investigator, PD Dr. Grégoire Wuerzner, MD, privat docent, MER, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Other Study IDs: 2017-00352
Record Dates: First submitted 2017-10-19; First posted 2017-10-24 (Actual); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: End Stage Renal Disease
Keywords: Blood pressure; Dialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HD - Hemodialysis: Patients with end stage renal disease treated with hemodialysis
- PD - Peritoneal dialysis: Patients with end stage renal disease treated with peritoneal dialysis

SUMMARY:
The objective of the current study is to evaluate the compliance to blood pressure measurements' recommendations in dialysis centers.

The idea is to address a questionnaire to physicians, head nurses and patients in order to probe the way to measure blood pressure. The objective is to face the theoretical guideline with what is effectively done.

DETAILED DESCRIPTION:
In dialysis center, blood pressure is measured as well as a vital sign than as a predictor of cardiovascular event. Accurate measurement of blood pressure is critical for making appropriate clinical decisions. Guidelines have been issued on standard blood pressure measurement procedure for the detection of hypertension and the follow-up of patients with hypertension. In hospital adherence to guidelines is low (Manzoli, Simonetti et al. 2012). Whether these guidelines are followed in dialysis patients is not known. Thus it would be of great interest to investigate the BP measurement procedures that are effectively applied in dialysis centers.

This project is an international survey across 10 dialysis centers. The current study is conducted on 10 physicians, 10 head nurses and 100 to 200 patients in Switzerland, in Europe and in the Mediterranean basin.

The adherence to BP measurement guidelines will be assessed thanks to two questionnaires of 20 items; one addressed to the patients and the other to the medical staff (clinicians and head nurses).

The project is scheduled to last a total of 4 months. Two months are dedicated to the presentation of the project, the recruitment as well as to the participation of the volunteers, and two months to the analysis.

The research project is carried out in accordance to the research plan and with principles enunciated in the current version of the Declaration of Helsinki (DoH), the Essentials of Good Epidemiological Practice issued by Public Health Schweiz (EGEP), the Swiss Law and Swiss regulatory authority's requirements as applicable.

ELIGIBILITY:
Inclusion Criteria:

* Dialysed patients (hemodialysis or peritoneal dialysis)

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from dialysis centers
Sampling Method: Non-Probability Sample
Enrollment: 192 (Estimated)
Dates: Start 2017-06-20 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Quality score | baseline
  To assess adherence to blood pressure measurement guidelines, a quality score is obtained from the surveys by assigning 1 point for each correct answer and 0 for the other one. The "perfect" and maximum score is 21. Higher scores indicate a better adherence to guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Grégoire Wuerzner, MD, Principal Investigator — Centre Hospitalier Universitaire Vaudois
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
it is planne to put IPD on zenodo Platform 1 year after publication